CLINICAL TRIAL: NCT05184647
Title: Total Splenectomy vs Partial Splenectomy in Non-malignant Hemoglobinopathies : Study Comparing the Effectiveness
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0712
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Splenectomy; Status
Keywords: Pediatrics; Non-malignant hemoglobinopathies; Comprative effectivness; Partial Splenectomy; Total Splenectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children under 18 years olds with total splenectomy for non Malignant hemoglobinopathie: Children under 18 years olds with total splenectomy for non Malignant hemoglobinopathie
- Children under 18 years olds with partial splenectomy for non Malignant hemoglobinopathie: Children under 18 years olds with partial splenectomy for non Malignant hemoglobinopathie

SUMMARY:
Partial splenectomy or total splenectomy are the two surgical treatment of non-malignant hemoglobinoptahie. The aim of this treatment is to decrease transfusion. The main risk is infectious in total splenectomy, that's why partial splenectomy was suggest. But the efficiency of partial splenectomy decrease over time and a totalisation could be mandatory.

ELIGIBILITY:
Inclusion criteria:

* Children between 0- 18 years olds
* Total or partial splenectomy
* Non malignant hémoglobinopathies

Exclusion criteria:

- Total or partial splenectomy outside of non malignant hemoglobinopathies

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children under 18 years olds with partial or total splenectomy for non malignant hemoglobinopathies
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-16 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Compared the effectiveness with the number of transfusion | Day 1
  Compared the effectiveness with the number of transfusion after the surgery between total and partial Febrile urinary tract infection was defined as a positive urine examination with a single bacteria with more than 10.5 cfu/mL and more than 10.4 leukocytes/ml associated with fever above 38.5°C and C-reactive protein (CRP) above 50 mg/

SECONDARY OUTCOMES:
Number of infectious event in total and partial splenectomy | Day 1
  Number of infectious event in total and partial splenectomy
number of totalisation in partial | Day 1
  number of totalisation in partial

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas KALFA, Study Director — University Hospital, Montpellier
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC